CLINICAL TRIAL: NCT05713175
Title: Effectiveness of Orthopaedic Treatment in Propulsive Metatarsalgia
Brief Title: Orthopaedic Treatment in Propulsive Metatarsalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tesis Doc Maria Ruiz-Ramos
Record Dates: First submitted 2022-10-05; First posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Metatarsalgia; Treatment; Foot; Foot Diseases; Orthopedic Disorder; Subluxation of Toe Joint; Toe Joint Deformity
Keywords: Metatarsalgia; Forefoot; Foot Diseases; Treatment
MeSH Terms: conditions — Metatarsalgia; Foot Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Groups Open Randomised Clinical Trial
Who Masked: Participant
Masking Description: The participant understands he is being part of a clinical trial but unknowns the treatment group he has been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EVA plantar orthosis (Active Comparator): Treatment consisting of a personalized plantar orthosis fabricated in 45º shore A hardness Ethyl Vinyl Acetate (EVA), which incorporates a 4mm heel rise and metatarsal dome placed proximal to the 2nd-3rd-4th metatarsal heads. No modifications applied to the patients' medial longitudinal arch.
  Interventions: Device: EVA plantar orthosis
- Polypropylene plantar orthosis (Active Comparator): Treatment consisting of a personalized plantar orthosis fabricated in 4mm polypropylene, which incorporates a 4mm heel rise and metatarsal dome placed proximal to the 2nd-3rd-4th metatarsal heads. No modifications applied to the patients' medial longitudinal arch.Orthosis fabricated following the inverted orthotic technique.
  Interventions: Device: Polypropylene plantar orthosis
- Fixtoe device (Active Comparator): Fixtoe device, simulating the metatarsophalangeal joint stabilization tape technique . Worn for one month, prior to definitive treatment.
  Interventions: Device: EVA plantar orthosis; Device: Polypropylene plantar orthosis; Device: Fixtoe device

INTERVENTIONS:
Device: EVA plantar orthosis — Treatment consisting of a personalized plantar orthosis fabricated in 45º shore A hardness Ethyl Vinyl Acetate (EVA), which incorporates a 4mm heel rise and metatarsal dome placed proximal to the 2nd-3rd-4th metatarsal heads. No modifications applied to the patients' medial longitudinal arch.
  Arms: EVA plantar orthosis; Fixtoe device
Device: Polypropylene plantar orthosis — Treatment consisting of a personalized plantar orthosis fabricated in 4mm polypropylene, which incorporates a 4mm heel rise and metatarsal dome placed proximal to the 2nd-3rd-4th metatarsal heads. No modifications applied to the patients' medial longitudinal arch.Orthosis fabricated following the inverted orthotic technique.
  Arms: Fixtoe device; Polypropylene plantar orthosis
Device: Fixtoe device — Fixtoe Device, simulating the metatarsophalangeal stabilization tape technique is worn for one month, prior to definitive treatment consisting of a personalized plantar orthosis.
  Arms: Fixtoe device

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two conservative orthopedic treatments in propulsive metatarsalgia.

The main question it aims to answer are:

* To compare the effectiveness of treatments on foot pain and functionality in subjects diagnosed with propulsive metatarsalgia.
* To determinate the influence of clinical and radiographical characteristics in pain improvement.

Participants will wear the treatment for 3 months . Researchers will compare polypropylene and EVA insoles and Fixtoe Device® to see if a foot pain improvement is achieved.

DETAILED DESCRIPTION:
Type of Study: Randomised Clinical Trial.

Aim: To compare the effect of orthopedic treatment on foot pain and functionality in subjects diagnosed with propulsive metatarsalgia.

Study Protocol Description:

Prior to the start of the study, a calculation of the sample size will be made using the GRANMO Sample Size Calculator, version .12 April 2012, with an error of 5%, assuming a confidence level of 95% and values of ß that establish an analysis power of 80%.

The study population will be randomly divided into two treatment groups, which, in turn, will be subdivided into two groups. Said randomization will be carried out using an online tool (www.randomization.com).

Treatment groups are:

* Group A: Treatment by custom insoles made of 4.5mm polypropylene, balanced in inversion 0-4º, MLA of the patient, 4mm-heel rise and metatarsal dome.
* Group A1: Treatment from the date of diagnosis until the start of insoles use (3 weeks) using the Fix-Toe® device.
* Group A2: Without orthopedic treatment from the date of diagnosis until the start of insoles use (3 weeks).
* Group B: Treatment by custom insoles made of 45º shore A E.V.A with the patient's MLA, 4mm- heel rise and metatarsal dome.
* Group B1: Treatment from the date of diagnosis until the start of insoles use (3 weeks) using the Fix-Toe® device.
* Group B2: Without orthopedic treatment from the date of diagnosis until the start of insoles use (3 weeks).

Visits protocol is as follows:

* Day 1: inclusion, clinical and radiographical evaluation. Pain questionnaires fulfillment.Treatment group allocation.
* Day 2 (3 weeks after Day 1): Pain questionnaires fulfillment. Starts insoles treatment.
* Day 3 (6 weeks after Day 2): Pain questionnaires fulfillment (telephone).
* Day 4 (6 weeks after Day 3): Pain questionnaires fulfillment. Clinical evaluation. End of study.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical pain in the 2nd or 3rd metatarsophalangeal joint (MTPJ)
* Positive Laschman's drawer test in 2nd or 3rd MTPJ. (CITA)
* Physical exploration revealing pain upon the palpation in plantar plate ( when cranial-caudal pressure was directly applied in the plantar aspect of the 2nd or 3rd MTPJ). (CITA)
* Availability of dorsal-plantar and lateral wheightbearing radiography of the affected foot.

Exclusion Criteria:

* Subjects with at least one of the following were excluded.
* Deformity of the 2nr or 3rd metatarsal head (MTH) (Freiberg's disease)
* Morton's neuroma and/or neuritic symptomatlogy y referred.
* Rigid claw or hammer toe (positive Kelikian test) whithin radiographic dislocation of 2nd or 3rd MTPJ. (CITA)
* Dermatological lesión plantar to 2nd or 3rd MTPJ (intractable plantar keratosis (IPK), foot ulcer, plantar wart, etc.)
* Neurological, methabolical, vascular or rheumatological not-controlled systemic disease with potential manifestations in foot and ankle.
* Previous history of foot or ankle surgery entailing limitations in mobility and/or alterations of the metatarsal parabola.
* Previous history of foot or ankle fracture
* Morpho-functional alteration of the lower limbs: clinical asymmetry greater than 10 mm and presence of asymmetric genu varus or valgus.
* Alterations of the cognitive state preventing to understand the objective of the study and guidelines to follow for their participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Foot Pain | Up to 20 weeks.
  Foot Pain measured using a 11-point VAS score. 0 is the lower (better) value and 10 is the higher (worst) value.
Foot Pain and Disability | Up to 20 weeks.
  Measured using the Foot Function Index (FFI-Sp) questionnaire (Spanish version). Higher values mean worse outcome and lower values mean better outcome.

SECONDARY OUTCOMES:
Demographic data: Age. | Day 1.
  Expressed in years
Demographic data: Gender | Day 1.
  Women or Men
Demographic data: Wheight | Day 1.
  Expressed in kilograms.
Demographic data: Height | Day 1.
  Expressed in centimetres.
Demographic data: Body Mass Index (BMI) | Day 1.
  Weight and Height will be combined to report BMI in kg/m^2
Demographic data: Adherence to treatment | Day 2, Day 3, Day 4.
  Good / Bad. Measured using a own questionnaire.
Demographic data: Time with symptoms. | Day 1.
  >12 months / 6-12 months / > 6 months / > 3 months
Foot clinical evaluation data: Toes deformity | Day 1.
  No deformity / Sagittal plane deformity / V sign
Foot clinical evaluation data: Paper pull-out test | Day 1, Day 2.
  No resistence / Medium resistence / Resistence
Foot clinical evaluation data: 1st metatarsophalangeal joint range of movement | Day 1, Day 4
  Expressed in degrees.
Foot clinical evaluation data: Medial column of the foot stiffness | Day 1.
  Low / Moderate/ High
Foot clinical evaluation data: Functional Hallux Limitus | Day 1.
  Yes / No. According to Functional Hallux Limitus test.
Foot clinical evaluation data: First ray mobility | Day 1.
  Dorsal > Plantar / Similar / Dorsal < Plantar
Foot clinical evaluation data: Lunge test | Day 1.
  Positive / Negative
Foot clinical evaluation data: Arch index | Day 1, Day 4.
  Expressed in degrees.
Foot clinical evaluation data: Navicular Drop Test | Day 1, Day 4.
  Expressed in centimetres.
Foot clinical evaluation data: Calcaneus relaxed standing position. | Day 1, Day 4.
  Expressed in degrees.
Foot clinical evaluation data: Subtalar joint axis orientation | Day 1.
  Medial / Neutral / Lateral
Radiographical data: HAV angle | Day 1.
  Expressed in degrees.
Radiographical data: 1st metatarsophalangeal joint osteoarthritis | Day 1.
  0/ 1/ 2/ 3/ 4
Metatarsal formula | Day 1.
  According to the length of the metatarsal bones.
Radiographical data: 2nd metatarsophalangeal joint angle | Day 1.
  Expressed in degrees.
Radiographical data: 3rd metatarsophalangeal joint angle | Day 1.
  Expressed in degrees.
Radiographical data: M1-M2 intermetatarsal angle | Day 1.
  Expressed in degrees.
Radiographical data: 2nd- 3rd metatarsophalangeal joint impingement | Day 1.
  Yes / No
Radiographical data: 2nd - 3rd metatatsophalangeal joint radiolucency. | Day 1.
  Yes / No
Radiographical data: Metatarsus primus elevatus | Day 1.
  Yes / No
Radiographical data: 1st cuneiform - 2nd metatarsal gap | Day 1.
  Expressed in centimetres.
Radiographical data: talar coverage angle | Day 1.
  Expressed in degrees.
Radiographical data: 1st cuneiform - 5th metatarsal distance | Day 1.
  Expressed in centimetres.
Radiographical data: Meary's line | Day 1.
  Dorsal / Plantar
Foot orthosis data: Metatarsal dome location in relation to central metatarsal heads | Day 4.
  Similar / Distal / Proximal
Foot orthosis data: Metatarsal dome location in relation to 1st metatarsal head | Day 4.
  Similar / Distal / Proximal
Foot orthosis data: Stability | Day 4.
  Yes / No
Foot orthosis data: Orthotic deformity test | Day 4.
  Yes / No

CONTACTS AND LOCATIONS:
Overall Officials: Ángel M Orejana-García, PhD, Study Director — Complutense University Madrid; Raúl J Molines-Barroso, PhD, Study Director — Complutense University Madrid; José Luis Lázaro-Martínez, PhD, Study Director — Complutense University Madrid; Maria Ruiz-Ramos, MSc, Principal Investigator — Complutense University Madrid
Locations (1):
- Clínica Universitaria de Podología Complutense University Madrid, Madrid, Spain